CLINICAL TRIAL: NCT07148284
Title: Characterization of EVs (Extracellular Vesicles)/miRNAs (microRNAs) From Human Follicular Fluid
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: ONZ-2024-0499; G096624N (Other Grant/Funding Number: FWO)
Record Dates: First submitted 2025-08-22; First posted 2025-08-29 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Extracellular Vesicles
Keywords: Extracellular vesicles; RNA sequencing
MeSH Terms: interventions — Sequence Analysis, RNA

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ≤ 32 years (Active Comparator)
  Interventions: Other: Isolation of EVs + RNA sequencing
- ≥ 38 years (Active Comparator)
  Interventions: Other: Isolation of EVs + RNA sequencing

INTERVENTIONS:
Other: Isolation of EVs + RNA sequencing — Isolation of EVs + RNA sequencing

SUMMARY:
* Background Extracellular vesicles (EVs) are membrane-bound vesicles found in all biological fluids. They contain various regulatory molecules, including microRNAs (miRNAs). It is hypothesized that EVs in human follicular fluid (the fluid surrounding the oocyte within the ovary) play a crucial role in oocyte development through these miRNAs.
* Research Question Is there a difference in miRNA expression in EVs in human follicular fluid based on the patient's age, the maturation stage of the corresponding oocyte, and/or the ploidy status of the resulting embryo (euploid in the case of a normal chromosome count vs. aneuploid in the case of an abnormal chromosome count)?
* Methodology This prospective study will include patients in two age groups (≥ 38 years vs. ≤ 32 years; 7 patients per group) undergoing an ICSI treatment (intracytoplasmic sperm injection) in combination with a coPGT-M treatment at Ghent University Hospital. PGT-M (pre-implantation genetic testing for monogenic disorders) is an IVF/ICSI procedure in which an embryo biopsy is performed on day 5 or 6 of embryo development to test for known genetic disorders that could be inherited from one or both parents. With the coPGT-M technology or comprehensive PGT-M, in addition to detecting known genetic defects, any additional chromosomal abnormalities in the embryo are also identified. An embryo is considered aneuploid if its chromosome number is abnormal.

For the participating patients, follicular fluid and plasma will be collected, and consent will be requested to store non-developing oocytes and embryos from the ICSI treatment.

Inclusion will take place on day 10 of ovarian stimulation if the patient meets the inclusion and exclusion criteria and at least 5 follicles are confirmed to be growing.

* Follicular Fluid (residual material): After oocyte retrieval, follicular fluid will be collected from 2-10 follicles per patient. EV isolation from this follicular fluid will be performed using the optimal technique determined in a preceding experiment (ID 18220, see 'Relations', comparison of 3 existing techniques to determine the optimal EV isolation technique from human follicular fluid). RNA extraction followed by miRNA sequencing will be used to assess differences in miRNA expression based on age (≤ 32 years vs. ≥ 38 years), oocyte maturation stage (mature vs. immature), and the ploidy status of the resulting embryo (euploid vs. aneuploid). In addition, the following hormone concentrations will be determined in the follicular fluid: estradiol, progesterone, follicle-stimulating hormone (FSH), and luteinizing hormone (LH).
* Plasma: For participating patients, an additional blood tube will be taken during each blood sample/infusion placement within the standard-of-care IVF/ICSI treatment from day 10 of ovarian stimulation until the day of oocyte retrieval. EV isolation and RNA extraction will be performed on plasma samples of the ovulation trigger day and oocyte retrieval day. MiRNA sequencing of these samples will be correlated with the miRNA expression of EVs in follicular fluid.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent.
* Oocyte retrieval planned for an coPGT-M ICSI trajectory at Ghent University Hospital.
* BMI 18,5-30 kg/m2.
* Normal karyotype of patient and partner.
* Ovarian stimulation protocol: PPOS (progestin-primed ovarian stimulation) with recombinant gonadotropins and GnRH agonist trigger.
* A minimum of 5 growing follicles during ovarian stimulation.

Exclusion Criteria:

* Diagnosis of endometriosis
* Diagnosis of PCOS according to Rotterdam criteria
* Poor ovarian responders according to Bologna criteria
* Severe male subfertility: semen concentration < 5 million/ml or TESE

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 14 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Differential miRNA expression based on the ploidy status of the resulting embryo | 6 months

SECONDARY OUTCOMES:
Differential miRNA expression based on the patient's age | 6 months
Differential miRNA expression based on the maturation stage of the corresponding oocyte | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Ghent University Hospital, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No